CLINICAL TRIAL: NCT00811213
Title: SASQT: SensAwake™ Sleep Quality Trial A Study to Test the Efficacy of the SensAwake™ Modification to Automatically Titrating Continuous Positive Airway Pressure to Reduce Wake After Sleep Onset in Patients With Moderate to Severe Obstructive Sleep Apnea.
Brief Title: SensAwake™ Sleep Quality Trial
Acronym: SASQT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Jessica Hayward Clinical Research Scientist, Fisher & Paykel Healthcare
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FP-08E-108
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Auto adjusting Continuous Postive Aiway Pressure (CPAP) Device with SensAwake technology enabled
  Interventions: Device: SleepStyle 200 Auto Series with SensAwake
- 2 (Active Comparator): Auto adjusting Continuous Postive Aiway Pressure (CPAP) Device with SensAwake technology disabled
  Interventions: Device: SleepStyle 200 Auto Series with out SensAwake

INTERVENTIONS:
Device: SleepStyle 200 Auto Series with SensAwake — Auto adjusting Continuous Postive Aiway Pressure (CPAP) Device with SensAwake technology enabled
  Arms: 1
Device: SleepStyle 200 Auto Series with out SensAwake — Auto adjusting Continuous Postive Aiway Pressure (CPAP) Device with SensAwake technology disabled
  Arms: 2

SUMMARY:
The SensAwake™ modification to the Fisher and Paykel automatically titrating positive airway pressure (APAP) device aims to sense whether the patient is awake via respiratory patterns that differentiate between sleep and wake. Upon sensing that the patient is awake the device is able to reduce positive airway pressure PAP aiming to improve patient comfort which should result in more consolidated sleep. This study will investigate Obstructive Sleep Apnea (OSA) and a automatically Adjusting Positive Airway Pressure (APAP) device with new technology called SensAwake™. This requires experimental confirmation in a randomised controlled trial. Double-blind randomised crossover trial comparing WASO on standard APAP with WASO using APAP modified by the addition of the SensAwake™ modification on consecutive nights in participants with moderate-to-severe OSA.

A total number of 45 participants will be recruited from an OSA population, aged 18-65. Participants will consist of male and female patients diagnosed with moderate-severe OSA (Apnea Hypopnea Index (AHI) greater than or equal to 15 per hour. Eligible participants, according to the protocol approved by the HREC, providing written informed consent will be enrolled into the study. Patients will be enrolled sequentially according to the randomisation list. Patients will be randomised to APAP or APAP with the addition of the SensAwake™ modification. The investigator and study staff will be blinded to the treatment of any participant.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years with moderate-to-severe OSA (Apnea Hypopnea index equal to or greater than 15 per hour).
* Epworth Sleepiness Scale (ESS) scores 0-15 inclusive (normal to moderately severe daytime sleepiness).
* Fluency in both written and spoken English.
* Do not have unstable psychiatric disease.
* No other significant sleep disorder.

Exclusion Criteria:

* Participants prescribed and fitted with any PAP device in the past 2 years.
* Unstable cardiovascular disease (untreated or resistant hypertension acceptable).
* Inability to tolerate CPAP due to nasal obstruction or claustrophobia as determined by the study investigator.
* Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results such as psychiatric disease, history of non compliance to medical regimens, or unwillingness to comply with study requirements.
* Participation in another clinical trial in the previous month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change in Wake After Sleep Onset (WASO) between treatment with standard APAP and APAP modified by the addition of the SensAwake™ modification | 1 Night

SECONDARY OUTCOMES:
Sleep Efficiency | 1 night
Percentage of Slow Wave Sleep | 1 night

CONTACTS AND LOCATIONS:
Overall Officials: Brendon Yee, MBChB, Principal Investigator — Woolcock Institute of Medical Research
Locations (1):
- Woolcock Institute of Medical Research, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Dungan GC 2nd, Marshall NS, Hoyos CM, Yee BJ, Grunstein RR. A randomized crossover trial of the effect of a novel method of pressure control (SensAwake) in automatic continuous positive airway pressure therapy to treat sleep disordered breathing. J Clin Sleep Med. 2011 Jun 15;7(3):261-7. doi: 10.5664/JCSM.1066. PMID 21677895
- See also: Study Site — http://www.woolcock.org.au/
- See also: Sponsor site — http://www.fphcare.co.nz/